CLINICAL TRIAL: NCT06215937
Title: Quantitative Sensory Testing and Central Sensitization in Endometriosis
Status: Recruiting | Type: Observational
Sponsor: BC Women's Hospital & Health Centre (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Paul Yong, Associate Professor, BC Women's Hospital & Health Centre
Other Study IDs: H22-02631
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis; Pain
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
Endometriosis is a gynecologic condition where there is growth of endometrial-like tissue outside the uterus, leading to severe pelvic pain. Despite conventional treatment, many patients experience persistent pelvic pain due to central sensitization (CS), where the central nervous system amplifies pain signals. Quantitative Sensory Testing (QST) enables objective testing of CS. However, there are several patient-reported questionnaires that have shown promising potential as subjective proxies of CS.

Therefore, in this study, our objective is to validate six patient-reported questionnaires as measures of CS by comparing them to each other and determining whether each questionnaire correlates with QST thresholds.

DETAILED DESCRIPTION:
Purpose: To validate the Central Sensitization Inventory (CSI), the Pain Sensitivity Questionnaire (PSQ), the Douleur Neuropathique 4 (DN4) questionnaire, the painDETECT (PD-Q) questionnaire, the Self Administered Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) and the Fibromyalgia (FM) Survey Score (FSS) as subjective proxies for detecting CS in cases of endometriosis.

Justificaiton: There has yet to be a direct comparison among these six questionnaires in endometriosis. Further research is needed to explore the overlap and effectiveness of these measures in the context of endometriosis and CS. Moreover, these six questionnaires have not been validated with quantitative sensory testing (QST) in endometriosis.Quantitative Sensory testing (QST) is an objective assessment tool for measuring CS. It quantifies the dynamic, altered modulation of nociceptive signals and allows for the objective testing of somatosensory function and central sensitization by applying various stimuli (such as pressure, pinprick, temperature etc.) to different body regions and recording pain thresholds (Rolke et al., 2006). Therefore, in this study, our objective is to compare the six patient-reported questionnaires to each other, and determine whether each questionnaire correlates with QST thresholds.

Primary Objective: Validate the CSI/PSQ/DN4/PD-Q/S-LANSS/FSS questionnaires as proxies for detecting CS in cases of endometriosis.

1. Examine the correlation between each questionnaire's scores with each other and the number of central sensitivity syndromes and other pelvic pain-related comorbidities (CSS) in patients with endometriosis.
2. Examine the association between questionnaire scores and the baseline QST thresholds in patients with endometriosis.

Secondary Objectives: Examine how the questionnaires and QST thresholds, correlate with pain severities, quality-of-life measured using the Endometriosis Health Profile (EHP-30) scores, demographic variables, as well as examination and surgical phenotyping of endometriosis.

Hypothesis: Higher scores on the CSI/PSQ/DN4/PD-Q/S-LANSS/FSS questionnaires will be associated with lower QST thresholds (as well as an increased number of CSS and other pelvic pain-related conditions) indicating greater central sensitization) in people with endometriosis

Research Design: This study is a cross-sectional correlational study, where all data points will be collected from participants at one point in time. The data collection process will include the collection of scores on six pain questionnaires (i.e.CSI, PSQ, DN4, PD-Q, S-LANSS and FSS) and threshold data from QST. All participants will be asked to complete the questionnaires. Depending on QST eligibility, determined during the screening assessment, and informed consent, a subgroup of participants will be asked to complete additional QST to obtain threshold data. The data analyses will focus on examining the relationships between each questionnaire and, for participants undertaking both the questionnaires and QST, the relationship between QST thresholds and each questionnaire.

Independent variables: Scores from the following questionnaires:

* CSI: CSI total score
* PSQ: PSQ minor score (avg. of scores from items 3,6,7,10,11,12,14) and the PSQ total score (avg. of scores from items 1,2,3,4,6,7,8,10,11,12,14,15,16)
* DN4: DN4 total score (sum of scores from items 1-7)
* PD-Q: PD-Q total score (sum of 7 sensory questions)
* S-LANSS: SLANSS total score
* FSS: FSS total score (WPI+ SS= SS) Main Outcome Variables: QST thresholds for assessment of CS PPT: avg. of duplicated PPT (kPa) at each test site VDT: avg. of VDT (Hz) at each test site MPT: avg. of duplicated MPT (NmN) at each test site MDT: avg. pain intensity rating on a 0-100' numerical rating scale (NRS) at each site SR- Fucntion: avg. pain intensity rating on a 0-100' numerical rating scale (NRS) at each site WUR: avg. of 5 WUR measurements (NmN) CPT: avg. of duplicated CPT (℃) at each test site CDT: avg of CDT (℃) at each test site HPT: avg. of duplicated HPT (℃) at each test site WDT: avg. of WDT (℃) at each test site CPM: avg. cearly CPM-effect and late CPM-effecthange in HPT (pain intensity on NRS)

Analysis of Data:All statistical analysis will be conducted using R or IBM SPSS, statistical software that allows for advanced data analysis, modelling, and visualization. For the primary analysis, we will conduct correlation analysis (Pearsons or Spearman's correlation) to assess the correlation, strength and direction of the associations between each questionnaire with each other and with other pelvic pain comorbidities (CSS). We will also examine the correlation/association between scores on each questionnaire and baseline QST thresholds. We will also determine lower QST thresholds correlate with an increasing number of CSS. For our secondary analysis, summary statistics, bivariate testing, T-tests, Mann-Whitney U test or Kruskal-Wallis tests will be conducted to determine the association between questionnaires and QST thresholds, and with various socioeconomic, demographic and anatomical phenotyping factors (e.g., endometriosis Stage, anatomic subtypes, histological confirmation, coexisting adenomyosis). We will also conduct correlation analysis to determine the association between pain severities and scores on the EHP-30. Regression analyses may be done with adjustments will be made for potential confounders (e.g. age, endometriosis stage and hormone therapy). All findings will be considered statistically significant at a threshold of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* New or re-referral appointment at the BC Women's Centre for Pelvic Pain and Endometriosis.
* Consented to be contacted for future research in the centre data registry (EPPIC NCT02911090; H16-00264).
* Surgically confirmed endometriosis, current imaging diagnosis, or current clinically suspected endometriosis diagnosed at the new or re-referral appointment as coded in the registry.
* 19 to 49 years old.
* Willing and committed to completing six questionnaires about pain.

QST specific criteria

• Willing and committed to QST testing.

Exclusion Criteria:

* Currently pregnant or breastfeeding.
* Post-menopausal.
* Does not speak English - Patients who do not speak English will be excluded to maintain the safety and well-being of the patient, as not understanding the test and process may harm the patient and reduce the validity of the results. We do not have research funding for a translator. Additionally, patients who require a translator are not typically included in the data registry and therefore are unlikely to be in our sample.

QST specific criteria

* Diabetes or neurological disease predisposing to neuropathic pain.
* Previous laparotomy (i.e. large abdominal incision)
* Physical trauma (ex., surgery, scaring) to heterotropic QST test site(s) (i.e. deltoid muscle in the shoulder, thenar eminence).

Ages: 19 Years to 49 Years | Sex: Female
Age Groups: Adult
Study Population: Individuals who have a new or re-referral appointment at the BC Women's Centre for Pelvic Pain and Endometriosis and who consented to the EPPIC registry (H16-00264).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization | Feb 1st 2023 - Jan 31st 2026
  Quantitative Sensory Testing thresholds for assessment of Central Sensitization

CONTACTS AND LOCATIONS:
Locations (1):
- BC Women's Hospital + Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No